CLINICAL TRIAL: NCT04191135
Title: An Open-label, Randomized, Phase 2/3 Study of Olaparib Plus Pembrolizumab Versus Chemotherapy Plus Pembrolizumab After Induction of Clinical Benefit With First-line Chemotherapy Plus Pembrolizumab in Participants With Locally Recurrent Inoperable or Metastatic Triple Negative Breast Cancer (TNBC) (KEYLYNK-009)
Brief Title: Study of Olaparib Plus Pembrolizumab Versus Chemotherapy Plus Pembrolizumab After Induction With First-Line Chemotherapy Plus Pembrolizumab in Triple Negative Breast Cancer (TNBC) (MK-7339-009/KEYLYNK-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7339-009; MK-7339-009 (Other: MSD); KEYLYNK-009 (Other: MSD); 195082 (Registry Identifier: JAPIC-CTI); 2022-500418-24-00 (Registry Identifier: EU CT); U1111-1275-8575 (Registry Identifier: UTN); 2019-001892-35 (EudraCT Number)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Programmed Cell Death Receptor 1 (PD-1, PD1); Programmed Cell Death Receptor Ligand 1 (PD-L1, PDL1); Programmed Cell Death Receptor Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; olaparib; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Olaparib (Experimental): This arm includes participants who randomized following completion of the induction period. After the induction period, participants received pembrolizumab 200 mg intravenously on Day 1 of each 21-day cycle plus olaparib 300 mg orally twice daily during the post-induction period.
  Interventions: Biological: Pembrolizumab; Drug: Olaparib
- Pembrolizumab + Carboplatin + Gemcitabine (Experimental): This arm includes participants who randomized following completion of the induction period. Participants continued to receive both carboplatin AUC 2 with gemcitabine 1000 mg/m^2 intravenously on Days 1 and 8 of each 21-day cycle in addition to pembrolizumab 200 mg intravenously on Day 1 of each 21-day cycle in the post-induction period.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Biological: Pembrolizumab — intravenous (IV) infusion
  Other Names: KEYTRUDA®; MK-3475
Drug: Olaparib — oral tablets
  Other Names: LYNPARZA®; MK-7339; AZD2281; KU-0059436
  Arms: Pembrolizumab + Olaparib
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
  Arms: Pembrolizumab + Carboplatin + Gemcitabine
Drug: Gemcitabine — IV infusion
  Other Names: GEMZAR®
  Arms: Pembrolizumab + Carboplatin + Gemcitabine

SUMMARY:
The purpose of this study is to compare the efficacy of olaparib (MK-7339) plus pembrolizumab (MK-3475) with chemotherapy plus pembrolizumab after induction with first-line chemotherapy plus pembrolizumab in triple negative breast cancer (TNBC). The primary hypotheses are:

1. Olaparib plus pembrolizumab is superior to chemotherapy plus pembrolizumab with respect to progression-free survival (PFS).
2. Olaparib plus pembrolizumab is superior to chemotherapy plus pembrolizumab with respect to overall survival (OS).

As of Amendment 3, study enrollment was discontinued. Participants who were receiving benefit from the study intervention could continue treatment until criteria for discontinuation are met. Participants who are on study treatment or in follow-up phase will no longer have tumor response assessments by BICR.

ELIGIBILITY:
Inclusion Criteria:

Induction Period:

* Has locally recurrent inoperable TNBC that has not previously been treated with chemotherapy and that cannot be treated with curative intent OR has metastatic TNBC that has not been previously treated with chemotherapy
* Has been treated with anthracycline and/or a taxane in the neoadjuvant/adjuvant setting, if they received systemic treatment in the neoadjuvant/adjuvant setting, unless anthracycline and/or taxane was contraindicated or not considered the best treatment option for the participant in the opinion of the treating physician
* Has measurable disease based on RECIST 1.1
* Has provided a recently obtained or archival (no more than 3 years old) core or excisional biopsy of a tumor lesion not previously irradiated
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 as assessed within 7 days prior to the start of induction study treatment
* Has a life expectancy ≥27 weeks from the day of first study treatment
* Demonstrate adequate organ function within 10 days prior to the start of study treatment
* A male participant must agree to be abstinent or use contraception and refrain from donating sperm during the intervention period and for at least the time needed to eliminate each study intervention (95 days for olaparib and chemotherapy; no requirement for pembrolizumab)
* A female participant must not be pregnant or breastfeeding and must agree to the following if is a woman of childbearing potential (WOCBP): have a negative pregnancy test within 24 hours before the start of study treatment and agree to be abstinent or use contraception and refrain from donating eggs (ova, oocytes) during the intervention period and for at least the time needed to eliminate each study intervention (180 days for olaparib and chemotherapy; 120 days for pembrolizumab)

Post-induction Period:

* Has received up to 6 cycles but not less than 4 cycles of induction therapy without permanently discontinuing from pembrolizumab or both carboplatin and gemcitabine
* Has achieved complete response (CR), partial response (PR), or stable disease (SD) based on RECIST 1.1 by Blinded Independent Central Review (BICR) at the Week 18 evaluation
* Is able to complete during post-induction at least the Cycle 1, Day 1 doses of olaparib and pembrolizumab or the Cycle 1, Day 1 doses of at least one of the chemotherapy agents being administered at the end of induction (carboplatin and/or gemcitabine) in addition to pembrolizumab
* Has ECOG performance status of 0 or 1, as assessed within 7 days prior to the start of post-induction study treatment
* Has no higher than Grade 1 toxicities related to induction therapy (excluding alopecia) prior to randomization

Exclusion Criteria:

Induction Period:

* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, cervical cancer in situ) that have undergone potentially curative therapy
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or has features suggestive of MDS/AML
* Has a history of (non-infectious) pneumonitis\interstitial lung disease that required steroids or current pneumonitis\interstitial lung disease
* Has active, or a history of, interstitial lung disease
* Has a known history of active tuberculosis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
* Has a history of class II-IV congestive heart failure or myocardial infarction within 6 months of first study treatment
* Has neuropathy ≥Grade 2
* Has not recovered (eg, to ≤Grade 1 or to baseline) from AEs due to a previously administered therapy
* Has a known history of hypersensitivity or allergy to pembrolizumab, olaparib and any of its components, and/or to any of the study chemotherapies (eg, carboplatin or gemcitabine) and any of their components
* Has severe hypersensitivity (≥Grade 3) to the study treatments and/or any of their excipients
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 180 days after the last dose of study treatment
* Is a WOCBP who has a positive urine pregnancy test within 24 hours prior to randomization or treatment allocation
* Has received prior therapy with either olaparib or any other poly adenosine diphosphate ribose polymerase (PARP) inhibitor
* Has received prior radiotherapy within 2 weeks of start of study treatment
* Has received colony-stimulating factors (eg, granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony stimulating factor [GM-CSF] or recombinant erythropoietin) within 2 weeks prior to the first dose of study treatment
* Has had an allogenic tissue/solid organ transplant.
* Has received previous allogenic bone marrow transplant or double umbilical cord transplantation (dUCBT)
* Has had major surgery within 2 weeks of starting study treatment or has not recovered from any effects of any major surgery
* Has received a live or live-attenuated vaccine within 30 days prior to first study treatment
* Is receiving any medication prohibited in combination with study chemotherapies unless medication was stopped within 7 days prior to first study treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T cell receptor (such as cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137) or has previously participated in a study evaluating pembrolizumab regardless of treatment received
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has presence of uncontrolled, potentially reversible cardiac conditions, as judged by the investigator
* Has a history or current evidence of any condition (eg, cytopenia, transfusion-dependent anemia, or thrombocytopenia), therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's involvement for the full duration of the study, or is not in the best interest of the participant to be involved, in the opinion of the treating investigator
* Is either unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (eg, gastrectomy, partial bowel obstruction, malabsorption)
* Is unlikely to comply with the study procedures, restrictions, and requirements of the study; as judged by the investigator

Post-induction Period:

* Has severe hypersensitivity (≥Grade 3) to the study treatments and/or any of their excipients
* Has permanently discontinued from both carboplatin and gemcitabine during induction due to toxicity
* Has permanently discontinued from pembrolizumab during induction due to toxicity
* Has received less than 4 cycles of chemotherapy plus pembrolizumab during induction
* Is currently receiving either strong or moderate inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study
* Is currently receiving either strong or moderate inducers of CYP3A4 that cannot be discontinued for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2025-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (122):
- United States (25):
  - Pacific Cancer Care ( Site 0142), Monterey, California
  - UCSF Helen Diller Family Comprehensive Cancer Center ( Site 0138), San Francisco, California
  - John Wayne Cancer Institute ( Site 0111), Santa Monica, California
  - St. Joseph Heritage Healthcare ( Site 0104), Santa Rosa, California
  - University of Miami Sylvester CC ( Site 0146), Miami, Florida
  - Georgia Cancer Center at Augusta University ( Site 0129), Augusta, Georgia
  - University of Chicago ( Site 0159), Chicago, Illinois
  - Massachusetts General Hospital ( Site 0155), Boston, Massachusetts
  - Henry Ford Health System ( Site 0103), Detroit, Michigan
  - Virginia Piper Cancer Institute ( Site 0157), Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center- Monmouth ( Site 0161), Middletown, New Jersey
  - MSKCC-Bergen ( Site 0162), Montvale, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack ( Site 0160), Commack, New York
  - Memorial Sloan-Kettering Cancer Center ( Site 0156), New York, New York
  - Mercy Clinic Oncology and Hematology ( Site 0110), Oklahoma City, Oklahoma
  - The Center For Cancer And Blood Disorders ( Site 0151), Fort Worth, Texas
  - Texas Oncology-New Braunfels ( Site 0168), New Braunfels, Texas
  - Texas Oncology-San Antonio Northeast ( Site 0165), San Antonio, Texas
  - Texas Oncology-San Antonio Medical Center ( Site 0158), San Antonio, Texas
  - Texas Oncology - San Antonio Stone Oak ( Site 0166), San Antonio, Texas
  - Renovatio Clinical ( Site 0117), The Woodlands, Texas
  - Virginia Oncology Associates ( Site 0163), Newport News, Virginia
  - Virginia Oncology Associates ( Site 0153), Norfolk, Virginia
  - Virginia Oncology Associates ( Site 0164), Virginia Beach, Virginia
  - YVMH dba Virginia Mason Memorial/North Star Lodge Cancer Center ( Site 0128), Yakima, Washington
- Canada (5):
  - Princess Margaret Cancer Centre ( Site 0005), Toronto, Ontario
  - CSSS de Laval- Hopital de la Cite de la Sante ( Site 0011), Laval, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0003), Montreal, Quebec
  - Jewish General Hospital ( Site 0010), Montreal, Quebec
  - McGill University Health Centre ( Site 0002), Montreal, Quebec
- Chile (5):
  - IC La Serena Research ( Site 0511), La Serena, Coquimbo Region
  - Fundacion Arturo Lopez Perez ( Site 0500), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0501), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0510), Temuco, Región de la Araucanía
  - Oncocentro ( Site 0502), Viña del Mar, Región de Valparaíso
- Colombia (6):
  - Fundacion Colombiana de Cancerologia Clinica Vida ( Site 0601), Medellín, Antioquia
  - Clinica de la Costa Ltda. ( Site 0600), Barranquilla, Atlántico
  - Organizacion Clinica Bonnadona-Prevenir S.A.S. ( Site 0609), Barranquilla, Atlántico
  - Oncomedica S.A. ( Site 0606), Montería, Departamento de Córdoba
  - Fundacion Valle del Lili ( Site 0602), Cali, Valle del Cauca Department
  - Hemato Oncologos S.A. ( Site 0603), Cali, Valle del Cauca Department
- France (12):
  - Centre Francois Baclesse ( Site 1012), Caen, Calvados
  - CHU-Jean Minjoz ( Site 1013), Besançon, Doubs
  - Institut Claudius Regaud IUCT Oncopole ( Site 1001), Toulouse, Haute-Garonne
  - Centre de Cancerologie du Grand Montpellier ( Site 1009), Montpellier, Languedoc-Roussillon
  - CHR-METZ-THIONVILLE - Hopital de Mercy ( Site 1007), Metz, Moselle
  - Centre Jean Perrin ( Site 1003), Clermont-Ferrand, Puy-de-Dome
  - Centre Leon Berard ( Site 1018), Lyon, Rhone
  - Centre Henri Becquerel ( Site 1020), Rouen, Seine-Maritime
  - CHU Amiens Hopital Sud ( Site 1023), Amiens, Somme
  - Institut Gustave Roussy ( Site 1010), Villejuif, Val-de-Marne
  - Institut Sainte Catherine ( Site 1026), Avignon, Vaucluse
  - Hôpital Saint-Louis ( Site 1025), Paris
- Germany (11):
  - Universitaetsklinikum Mannheim GmbH ( Site 1213), Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen ( Site 1201), Erlangen, Bavaria
  - Klinik und Poliklinik fuer Frauenheilkunde und Geburtshilfe ( Site 1200), Munich, Bavaria
  - Hochwaldkrankenhaus Bad Nauheim ( Site 1211), Bad Nauheim, Hesse
  - Sana Klinikum Offenbach Klinik fuer Gynakologie und Geburtshilfe ( Site 1206), Offenbach, Hesse
  - Gynaekologisch-onkologische Praxis Hannover ( Site 1207), Hanover, Lower Saxony
  - Gynaekologisches Zentrum-Schwerpunkt Gyn. Onkologie ( Site 1205), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum AoeR Duesseldorf ( Site 1210), Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte ( Site 1215), Essen, North Rhine-Westphalia
  - Frauenklinik St. Louise ( Site 1216), Paderborn, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus ( Site 1203), Dresden, Saxony
- Hungary (7):
  - Pecsi Tudomanyegyetem Klinikai Kozpont ( Site 1607), Pécs, Baranya
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 1608), Kecskemét, Bács-Kiskun county
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 1601), Szolnok, Jász-Nagykun-Szolnok
  - Zala Megyei Szent Rafael Korhaz ( Site 1605), Zalaegerszeg, Zala County
  - Orszagos Onkologiai Intezet ( Site 1602), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 1600), Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 1604), Kaposvár
- Ireland (2):
  - Cork University Hospital ( Site 0902), Cork
  - St Vincents University Hospital ( Site 0900), Dublin
- Japan (5):
  - Aichi Cancer Center Hospital ( Site 2202), Nagoya, Aichi-ken
  - Hyogo College of Medicine Hospital ( Site 2203), Nishinomiya, Hyōgo
  - Fukushima Medical University Hospital ( Site 2201), Fukushima
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2204), Hiroshima
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research (Site 2200), Osaka
- Poland (6):
  - Pleszewskie Centrum Medyczne w Pleszewie Sp. z o.o. ( Site 1909), Pleszew, Greater Poland Voivodeship
  - Pratia MCM Krakow ( Site 1919), Krakow, Lesser Poland Voivodeship
  - Regionalny Szpital Specjalistyczny Latawiec ( Site 1917), Swidnica, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (Site 1908), Warsaw, Masovian Voivodeship
  - Szpital Morski im. PCK. Szpitale Pomorskie Sp. Z o.o ( Site 1913), Gdynia, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 1912), Gliwice, Silesian Voivodeship
- South Korea (9):
  - National Cancer Center ( Site 2406), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 2409), Seongnam-si, Kyonggi-do
  - Ajou University Hospital ( Site 2407), Suwon, Kyonggi-do
  - Kyungpook National University Chilgok Hospital ( Site 2402), Daegu, Taegu-Kwangyokshi
  - Gachon University Gil Medical Center ( Site 2408), Incheon
  - Seoul National University Hospital ( Site 2403), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2401), Seoul
  - Asan Medical Center ( Site 2404), Seoul
  - Samsung Medical Center ( Site 2405), Seoul
- Spain (6):
  - Hospital Universitario Reina Sofia ( Site 0705), Córdoba, Andalusia
  - Hospital General Arnau de Vilanova de Valencia ( Site 0706), Valencia, Valenciana, Comunitat
  - Instituto Oncologico Baselga.Hospital Quiron. ( Site 0707), Barcelona
  - Hospital Universitari Vall d Hebron ( Site 0701), Barcelona
  - Hospital Clinic I Provincial de Barcelona ( Site 0702), Barcelona
  - Clinica Universitaria Navarra - Madrid ( Site 0700), Madrid
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital ( Site 2304), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 2303), Tainan
  - MacKay Memorial Hospital ( Site 2301), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 2300), Taipei
  - China Medical University Hospital ( Site 2302), Taipei
- Ukraine (12):
  - Chernihiv Medical Center of Modern Oncology ( Site 1520), Chernihiv, Chernihiv Oblast
  - Dnipropetrovsk City Multidiscipline Clinical Hosp. 4 of DRC ( Site 1502), Dnipro, Dnipropetrovsk Oblast
  - CI Krivorizhskiy oncology dispensery ( Site 1504), Kryviy Rih, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 1506), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 1508), Kharkiv, Kharkivs’ka Oblast’
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 1512), Kharkiv, Kharkivs’ka Oblast’
  - SI-Zaytsev institute of general and urgent surgery-NAMS ( Site 1518), Kharkiv, Kharkivs’ka Oblast’
  - Medical Centre Consilium Medical ( Site 1514), Kyiv, Kyivska Oblast
  - Medical center of the Limited Liability Company Yulis ( Site 1517), Zaporizhzhia, Zaporizhzhia Oblast
  - Medical Centre LLC Oncolife ( Site 1510), Zaporizhzhya, Zaporizhzhia Oblast
  - Zhytomyr Regional Oncology Center ( Site 1515), Zhytomyr, Zhytomyr Oblast
  - Medical Center Verum ( Site 1501), Kyiv
- United Kingdom (6):
  - Raigmore Hospital ( Site 0915), Inverness, Highland
  - Blackpool Victoria Hospital ( Site 0921), Blackpool, Lancashire
  - Barts Health NHS Trust ( Site 0912), London, London, City of
  - North West Cancer Centre ( Site 0922), Londonderry, London, City of
  - Musgrove Park Hospital ( Site 0918), Taunton, Somerset
  - The Christie NHS Foundation Trust ( Site 0914), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26195&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment: Participants receive both carboplatin Area Under The Curve (AUC) 2 with gemcitabine 1000 mg/m^2 intravenously on Days 1 and 8 of each 21-day cycle plus pembrolizumab 200 mg intravenously on Day 1 of each 21-day cycle during the induction period for 4-6 cycles. Participants may then randomize to one of the blinded treatment arms.
Period: Induction Treatment
Arm/Group | Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Started | 462 | 0 | 0
Treated | 460 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 462 | 0 | 0
Not completed — Not Treated | 2 | 0 | 0
Not completed — Ongoing to Blinded Treatment Period | 271 | 0 | 0
Not completed — Adverse Event | 25 | 0 | 0
Not completed — Clinical Progression | 8 | 0 | 0
Not completed — Excluded Medication | 1 | 0 | 0
Not completed — Failure to Meet Continuation Criteria | 2 | 0 | 0
Not completed — Failure to Meet Randomization Criteria | 2 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Progressive Disease | 135 | 0 | 0
Not completed — Protocol Violation | 10 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Period: Randomized Treatment
Arm/Group | Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Started | 0 | 135 (Per protocol, not all participants from the induction period continued into the randomized treatment period.) | 136 (Per protocol, not all participants from the induction period continued into the randomized treatment period.)
Treated | 0 | 135 | 133
Completed | 0 | 0 | 0
Not Completed | 0 | 135 | 136
Not completed — Death | 0 | 50 | 54
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Ongoing in Trial | 0 | 83 | 81

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment: Participants receive both carboplatin Area Under The Curve (AUC) 2 with gemcitabine 1000 mg/m^2 intravenously on Days 1 and 8 of each 21-day cycle plus pembrolizumab 200 mg intravenously on Day 1 of each 21-day cycle during the induction period for 4-6 cycles. These participants did not randomize to a post-induction arm.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine | Total
Number analyzed (Participants) | 189 | 135 | 136 | 460
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (12.7) | 53.9 (12.0) | 52.9 (12.5) | 53.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 135 | 136 | 459
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 33 | 19 | 78
  Not Hispanic or Latino | 137 | 79 | 102 | 318
  Unknown or Not Reported | 26 | 23 | 15 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 2 | 5
  Asian | 39 | 29 | 30 | 98
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 6 | 5 | 2 | 13
  White | 112 | 70 | 84 | 266
  More than one race | 7 | 14 | 7 | 28
  Unknown or Not Reported | 21 | 17 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR), or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters (SOD) of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: The analysis population included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 136
Months | 5.5 [4.2 to 8.3] | 5.6 [4.3 to 6.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.4556, Log Rank — One-sided p-value based on log-rank test stratified by response to the induction therapy (CR/PR versus SD), tumor PD-L1 status (CPS ≥1 vs CPS <1) and BRCA Status (BRCAm versus wild type BRCA gene); Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.72 to 1.33] — Estimate via stratified Cox model with Efron's handling method with treatment as a covariate stratified by response to the induction therapy (CR/PR versus SD), tumor PD-L1 status (CPS ≥1 vs CPS <1) and BRCA Status (BRCAm versus wild type BRCA gene)

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: The analysis population included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 136
Months | 25.1 [18.3 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 23.4 [15.8 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.3903, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.64 to 1.40] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Progression-Free Survival (PFS) in Participants With Programmed Cell Death-Ligand 1 (PD-L1) Positive Tumors With a Combined Positive Score (CPS) ≥10
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR), or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters (SOD) of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Only participants with a CPS ≥10 were included in this analysis. PFS is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: The analysis populations included all randomized participants with a CPS ≥10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 65 | 65
Months | 5.7 [2.9 to 13.9] | 5.7 [3.8 to 7.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Other; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.59 to 1.43] — Estimate based on stratified Cox model with Efron's method of tie handling with treatment as a covariate stratified by response to the induction therapy (CR or PR versus SD) and BRCA status (BRCAm versus BRCAwt)

4. Secondary Outcome: Overall Survival (OS) in Participants With PD-L1 Positive Tumors With a CPS ≥10
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Only participants with a CPS ≥10 were included in this analysis.
Time Frame: Up to approximately 29 months
Population: The analysis population included all randomized participants with a CPS ≥10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 65 | 65
Months | NA [17.0 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [15.5 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Other; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.53 to 1.76] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: PFS in Participants With Breast Cancer Susceptibility Gene Mutation (BRCAm) Tumors
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR), or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters (SOD) of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Only participants with BRCAm-positive tumors were included in this analysis. PFS is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: The analysis population included all randomized participants with BRCAm tumors
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Months | 12.4 [8.3 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 8.4 [5.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Other; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.33 to 1.48] — Estimate based on stratified Cox model with Efron's method of tie handling with treatment as a covariate stratified by response to the induction therapy (CR or PR versus SD) and tumor PD-L1 status (CPS≥1 vs CPS<1)

6. Secondary Outcome: OS in Participants With BRCAm Tumors
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Only participants with BRCAm-positive tumors were included in this analysis.
Time Frame: Up to approximately 29 months
Population: The analysis population included all randomized participants with BRCAm tumors
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Months | NA [17.1 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 23.4 [17.3 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.28 to 2.37] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline in Health-Related Quality-of-Life (QoL) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Items 29 and 30 Combined Score
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were each scored on a 7-point scale (1=Very Poor to 7=Excellent), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Change from baseline in EORTC QLQ-C30 Items 29 and 30 combined scores was calculated based on a constrained longitudinal data analysis (cLDA) model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1) and BRCA status at randomization (BRCAm vs. BRCAwt)) as covariates.
Time Frame: Baseline and week 18
Population: The analysis population included all randomized participants who received ≥1 dose of study treatment and who completed at least one assessment for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Score on a Scale | -5.82 [-9.03 to -2.61] | -2.54 [-5.71 to 0.64]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.1430, cLDA; cLDA model with PRO scores as the response variable with covariates for treatment by time interaction, stratification factors as covariates; Difference in Least Squares Means = -3.28, 95% CI 2-sided [-7.69 to 1.12]

8. Secondary Outcome: Change From Baseline in Physical Functioning Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Items 1- 5 Score
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. The change from baseline in physical functioning (EORTC QLQ-C30 Items 1-5) score was calculated based on a cLDA model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1) and BRCA status at randomization (BRCAm vs. BRCAwt)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Score on a Scale | -2.86 [-6.29 to 0.57] | -2.69 [-6.09 to 0.70]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.9454, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = -0.16, 95% CI 2-sided [-4.89 to 4.56]

9. Secondary Outcome: Change From Baseline in Emotional Functioning Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Items 21-24 Score
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 4 questions about their emotional functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Change from baseline in emotional functioning (EORTC QLQ-C30 Items 21-24) score was calculated based on a cLDA model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1) and BRCA status at randomization (BRCAm vs. BRCAwt)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Score on a Scale | -0.46 [-4.30 to 3.38] | -2.53 [-6.32 to 1.25]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.4351, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = 2.08, 95% CI 2-sided [-3.16 to 7.31]

10. Secondary Outcome: Change From Baseline in Systemic Therapy Side Effects Using the European Organization for Research and Treatment of Cancer Breast Cancer-Specific QoL Questionnaire (EORTC QLQ-BR23) Items 1-4, 6, 7, and 8 Score
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30, consisting of functional scales (body image, sexual enjoyment, sexual functioning, future perspective) and symptom scales (systemic therapy side effects, upset by hair loss, arm symptoms, breast symptoms). Participant responses to 7 questions about their systemic therapy side effects are scored on a 4-point scale (1=Not at All, 4=Very Much). Using linear transformation, raw scores are standardized, so scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in systemic therapy side effects (EORTC QLQ-BR23 Items 1-4, 6, 7, and 8) score was calculated based on a cLDA model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1) and BRCA status at randomization (BRCAm vs. BRCAwt)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Score on a Scale | -0.91 [-3.27 to 1.44] | -1.84 [-4.17 to 0.48]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.5588, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = 0.93, 95% CI 2-sided [-2.20 to 4.06]

11. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score on the European Quality of Life 5-dimension, 5-level Questionnaire (EQ-5D-5L)
Description: The EQ-5D-5L is a questionnaire developed to assess health-related outcomes. The VAS is a component of the EQ-5D-5L that asks participants to rate their overall health on a vertical visual analogue scale, with the scale's ends labelled 'The best health you can imagine' (equivalent to a score of 0) and 'The worst health you can imagine' (equivalent to a score of 100). The change from baseline in VAS score was calculated based on a cLDA model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1) and BRCA status at randomization (BRCAm vs. BRCAwt)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Score on a Scale | -2.74 [-5.36 to -0.12] | -2.37 [-4.97 to 0.24]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.8408, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = -0.37, 95% CI 2-sided [-4.03 to 3.28]

12. Secondary Outcome: Change From Baseline in Health-Related QoL Using the EORTC QLQ-C30 Items 29 and 30 Combined Score in Participants With Breast Cancer Susceptibility Gene Mutation (BRCAm) Tumors
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were each scored on a 7-point scale (1=Very Poor to 7=Excellent), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. The change from baseline in EORTC QLQ-C30 Items 29 and 30 scores was calculated based on a constrained longitudinal data analysis (cLDA) model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), and baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1)) as covariates.
Time Frame: Baseline and up to 18 weeks
Population: The analysis population included all randomized participants with BRCAm tumors, who received ≥1 dose of study treatment and who completed at least one assessment for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Score on a Scale | -4.85 [-12.43 to 2.73] | -3.51 [-11.17 to 4.15]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.7950, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = -1.34, 95% CI 2-sided [-11.63 to 8.95]

13. Secondary Outcome: Change From Baseline in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score in Participants With BRCAm Tumors
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. The change from baseline in physical functioning (EORTC QLQ-C30 Items 1-5) score was calculated based on a constrained longitudinal data analysis (cLDA) model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), and baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Score on a Scale | 4.12 [-0.68 to 8.92] | -0.70 [-5.62 to 4.21]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.1597, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = 4.82, 95% CI 2-sided [-1.97 to 11.62]

14. Secondary Outcome: Change From Baseline in Emotional Functioning Using the EORTC QLQ-C30 Items 21-24 Score in Participants With BRCAm Tumors
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 4 questions about their emotional functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. The change from baseline in emotional functioning (EORTC QLQ-C30 Items 21-24) score was calculated based on a cLDA model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), and baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Score on a Scale | -1.50 [-8.41 to 5.41] | -4.02 [-11.15 to 3.11]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.6138, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = 2.52, 95% CI 2-sided [-7.45 to 12.49]

15. Secondary Outcome: Change From Baseline in Systemic Therapy Side Effects Using the EORTC QLQ-BR23 Items 1-4, 6, 7, and 8 Score in Participants With BRCAm Tumors
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30, consisting of functional scales (body image, sexual enjoyment, sexual functioning, future perspective) and symptom scales (systemic therapy side effects, upset by hair loss, arm symptoms, breast symptoms). Participant responses to 7 questions about their systemic therapy side effects are scored on a 4-point scale (1=Not at All, 4=Very Much). Using linear transformation, raw scores are standardized, so scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in systemic therapy side effects (EORTC QLQ-BR23 Items 1-4, 6, 7, and 8) score was calculated based on a cLDA model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), and baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Score on a Scale | -4.27 [-8.27 to -0.27] | -2.67 [-6.77 to 1.43]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.5567, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = -1.60, 95% CI 2-sided [-7.02 to 3.83]

16. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score on the EQ-5D-5L in Participants With BRCAm Tumors
Description: The EQ-5D-5L is a questionnaire developed to assess health-related outcomes. The VAS is a component of the EQ-5D-5L that asks participants to rate their overall health on a vertical visual analogue scale, with the scale's ends labelled 'The best health you can imagine' (equivalent to a score of 0) and 'The worst health you can imagine' (equivalent to a score of 100). The change from baseline in VAS score was calculated based on a cLDA model with scores as response variable with covariates for treatment by time interaction, stratification factors (response at randomization (CR/PR vs. SD), and baseline CPS for PD-L1 expression (PD-L1 CPS<1 vs. PD-L1 CPS≥1)) as covariates.
Time Frame: Baseline and week 18
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Score on a Scale | 1.73 [-3.08 to 6.54] | -3.83 [-8.77 to 1.11]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.1050, cLDA; [statistical method as in outcome 7, analysis 1]; Difference in Least Squares Means = 5.56, 95% CI 2-sided [-1.20 to 12.32]

17. Secondary Outcome: Time to Deterioration (TTD) in Health-Related QoL Using the EORTC QLQ-C30 Items 29 and 30 Score
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were each scored on a 7-point scale (1=Very Poor to 7=Excellent), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. TTD was defined as the time from baseline to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in Items 29 and 30 scale scores. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Baseline and up to approximately 29 months
Population: The analysis population included all randomized participants who received ≥1 dose of study treatment and who completed the baseline assessment for this outcome.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Months | 10.3 [4.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [13.2 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.00676, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 1.78, 95% CI 2-sided [1.16 to 2.71] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: TTD in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. TTD was defined as the time from baseline to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in physical functioning Items 1 to 5 scale scores. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.96425, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.61 to 1.69] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: TTD in Emotional Functioning Using the EORTC QLQ-C30 Items 21-24 Score
Description: EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to 4 questions about their emotional functioning are scored on a 4-point scale (1=Not at All to 4=Very Much), then summed. Summed raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. TTD was defined as the time from baseline to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in emotional functioning Items 21-24 scale scores. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 132
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [14.5 to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.74965, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.69 to 1.71] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: TTD in Systemic Therapy Side Effects Using the EORTC QLQ-BR23 Items 1-4, 6, 7, and 8 Score
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective) and four symptom scales (systemic therapy side effects, upset by hair loss, arm symptoms, breast symptoms). Participant responses to 7 questions about their systemic therapy side effects are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. TTD was defined as the time from baseline to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in systemic therapy side effects Items 1-4, 6, 7 and 8 scale scores. TTD is reported based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 29 months
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 134 | 132
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.10502, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 1.76, 95% CI 2-sided [0.88 to 3.53] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: TTD in Health-Related QoL Using the EORTC QLQ-C30 Items 29 and 30 Score in Participants With Breast Cancer Susceptibility Gene Mutation (BRCAm) Tumors
Description: as for outcome 17
Time Frame: Baseline and up to approximately 29 months
Population: The analysis population included all randomized participants with BRCAm tumors, who received ≥1 dose of study treatment and who completed the baseline assessment for this outcome.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Months | 7.9 [3.7 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [3.5 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.50190, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.57 to 3.00] — Estimate via stratified Cox model with Efron's handling method with treatment as a covariate stratified by response to the induction therapy (CR/PR versus SD), and tumor PD-L1 status (CPS ≥1 vs CPS <1)

22. Secondary Outcome: TTD in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score in Participants With BRCAm Tumors
Description: as for outcome 18
Time Frame: Up to approximately 29 months
Population: as for outcome 21
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Months | NA [10.4 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.47384, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.24 to 1.97] — [estimate comment as in outcome 21, analysis 1]

23. Secondary Outcome: TTD in Emotional Functioning Using the EORTC QLQ-C30 Items 21-24 Score in Participants With BRCAm Tumors
Description: as for outcome 19
Time Frame: Up to approximately 29 months
Population: as for outcome 21
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Months | NA [7.9 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [15.4 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.81463, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.33 to 2.38] — [estimate comment as in outcome 21, analysis 1]

24. Secondary Outcome: TTD in Systemic Therapy Side Effects Using the EORTC QLQ-BR23 Items 1-4, 6, 7, and 8 Score in Participants With BRCAm Tumors
Description: as for outcome 20
Time Frame: Up to approximately 29 months
Population: as for outcome 21
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 29 | 30
Months | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, lower limit, and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib vs Pembrolizumab + Carboplatin + Gemcitabine; Test type: Superiority; p = 0.67255, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.24 to 8.82] — [estimate comment as in outcome 21, analysis 1]

25. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience at least 1 AE is presented.
Time Frame: Up to approximately 29 months
Population: The analysis population included all randomized participants who received ≥1 dose of study drug and who had at least 1 laboratory or vital sign measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 133
Participants | 126 | 130

26. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 29 months
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 135 | 133
Participants | 15 | 28

ADVERSE EVENTS:
Time Frame: Up to approximately 29 months
Description: Mortality includes all enrolled participants regardless of treatment status. AEs include all participants who received ≥1 dose of study drug, counted in the latest arm for which a participant received drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs.
Arm/Group | Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment | Pembrolizumab + Olaparib | Pembrolizumab + Carboplatin + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 124/460 | 50/135 | 54/136
Serious Adverse Events (participants affected / at risk) | 80/460 | 35/135 | 32/133
Other Adverse Events (participants affected / at risk) | 456/460 | 121/135 | 128/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment (N=460) | Pembrolizumab + Olaparib (N=135) | Pembrolizumab + Carboplatin + Gemcitabine (N=133)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 2 (3) | 2 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis noninfective (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (5) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Carboplatin + Gemcitabine Induction Treatment (N=460) | Pembrolizumab + Olaparib (N=135) | Pembrolizumab + Carboplatin + Gemcitabine (N=133)
Anaemia (Blood and lymphatic system disorders) | 274 (361) | 54 (75) | 69 (121)
Leukopenia (Blood and lymphatic system disorders) | 84 (179) | 16 (31) | 23 (65)
Lymphopenia (Blood and lymphatic system disorders) | 23 (37) | 11 (20) | 5 (18)
Neutropenia (Blood and lymphatic system disorders) | 218 (485) | 28 (54) | 55 (187)
Thrombocytopenia (Blood and lymphatic system disorders) | 133 (236) | 22 (30) | 41 (148)
Hyperthyroidism (Endocrine disorders) | 25 (25) | 1 (1) | 3 (3)
Hypothyroidism (Endocrine disorders) | 53 (53) | 13 (14) | 12 (12)
Abdominal pain (Gastrointestinal disorders) | 27 (31) | 12 (17) | 8 (9)
Abdominal pain upper (Gastrointestinal disorders) | 29 (34) | 5 (5) | 6 (7)
Constipation (Gastrointestinal disorders) | 141 (171) | 14 (14) | 13 (17)
Diarrhoea (Gastrointestinal disorders) | 66 (84) | 23 (30) | 22 (30)
Dyspepsia (Gastrointestinal disorders) | 29 (32) | 8 (8) | 7 (16)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 (19) | 7 (8) | 7 (10)
Nausea (Gastrointestinal disorders) | 207 (324) | 51 (59) | 36 (57)
Stomatitis (Gastrointestinal disorders) | 22 (27) | 8 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 83 (124) | 19 (25) | 22 (34)
Asthenia (General disorders) | 102 (142) | 22 (24) | 25 (36)
Fatigue (General disorders) | 124 (160) | 22 (25) | 23 (29)
Influenza like illness (General disorders) | 9 (13) | 8 (8) | 6 (8)
Pyrexia (General disorders) | 50 (62) | 11 (12) | 16 (32)
COVID-19 (Infections and infestations) | 11 (11) | 12 (12) | 18 (19)
Alanine aminotransferase increased (Investigations) | 162 (208) | 8 (8) | 32 (57)
Aspartate aminotransferase increased (Investigations) | 136 (173) | 10 (12) | 29 (47)
Blood alkaline phosphatase increased (Investigations) | 26 (30) | 5 (6) | 7 (11)
Blood creatinine increased (Investigations) | 3 (3) | 7 (10) | 5 (5)
Blood lactate dehydrogenase increased (Investigations) | 26 (28) | 5 (6) | 11 (15)
Lymphocyte count decreased (Investigations) | 26 (46) | 12 (27) | 11 (31)
Neutrophil count decreased (Investigations) | 141 (298) | 18 (33) | 42 (183)
Platelet count decreased (Investigations) | 95 (158) | 16 (22) | 36 (101)
White blood cell count decreased (Investigations) | 71 (149) | 14 (29) | 28 (78)
Decreased appetite (Metabolism and nutrition disorders) | 61 (70) | 24 (25) | 10 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 19 (20) | 7 (7) | 3 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (19) | 11 (14) | 9 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 (23) | 8 (11) | 12 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 (52) | 12 (15) | 22 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (31) | 15 (20) | 12 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 37 (44) | 7 (8) | 10 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (24) | 8 (8) | 10 (10)
Dizziness (Nervous system disorders) | 24 (29) | 6 (7) | 11 (13)
Dysgeusia (Nervous system disorders) | 29 (29) | 8 (10) | 2 (2)
Headache (Nervous system disorders) | 95 (129) | 28 (31) | 35 (52)
Neuropathy peripheral (Nervous system disorders) | 14 (14) | 3 (3) | 7 (7)
Anxiety (Psychiatric disorders) | 12 (12) | 10 (10) | 2 (2)
Insomnia (Psychiatric disorders) | 22 (25) | 7 (7) | 9 (10)
Breast pain (Reproductive system and breast disorders) | 14 (17) | 3 (3) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (34) | 10 (10) | 13 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 (36) | 5 (6) | 10 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0) | 7 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 55 (55) | 4 (4) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 45 (49) | 7 (7) | 9 (11)
Rash (Skin and subcutaneous tissue disorders) | 60 (66) | 5 (5) | 16 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 26 (32) | 3 (5) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04191135/Prot_SAP_000.pdf